CLINICAL TRIAL: NCT06681636
Title: A Non-inferiority Study Comparing the Immunogenicity of a Standard or an Extended Three-dose Nonavalent Human Papillomavirus Vaccine Schedule Between High-risk Women Aged 18-26 Years and Age-matched Women in the General Population
Brief Title: Effector and Memory Immune Responses to HPV Vaccination in Vietnamese Women Post Virus Exposure
Acronym: HPV9vxFSW
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Collaborators: Murdoch Childrens Research Institute (Other); CENTER FOR SUPPORTING COMMUNITY DEVELOPMENT INITIATIVES (Unknown); Hai Phong Center for Disease Control (Other Government)
Responsible Party: Principal Investigator, Nguyen Van Trang, Acting Manager, Center for Biomedical Researches, National Institute of Hygiene and Epidemiology, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HPV9-VINIF2427
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: HPV Infection; Cervical Cancer; Anogenital Cancer; Anogenital Warts
Keywords: human papillomavirus; HPV vaccine; Vietnam; Female sex workers; immunogenicity; protection; extended schedule; HPV infection; cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants (FSW groups) will be randomly assigned to either of the vaccine schedules and will be given IDs. The link between participant IDs and vaccine groups are only known by Investigator.
  Barcodes will be used for samples and no personal identification nor participant ID is allowed in the samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 FSW (Experimental): 100 FSWs aged 18-26 years receiving 3 doses of Gardasil-9 vaccine at 0-6-18 months
  Interventions: Biological: Human papillomavirus 9-valent vaccine, Recombinant
- Group 2 non-FSW (Active Comparator): 100 non-FSW aged 18-26 years receiving 3 doses of Gardasil-9 vaccine at 0-6-18 months
  Interventions: Biological: Human papillomavirus 9-valent vaccine, Recombinant
- Group 3 FSW (Active Comparator): 100 FSW aged 18-26 years receiving 3 doses of Gardasil-9 vaccine at 0-2-6 months
  Interventions: Biological: Human papillomavirus 9-valent vaccine, Recombinant

INTERVENTIONS:
Biological: Human papillomavirus 9-valent vaccine, Recombinant — HPV vaccine manufactured by MSD consisted of 9HPV types: 6,11,16,18,31,33, 45, 52,58
  Other Names: Gardasil 9

SUMMARY:
A Study to evaluate if the 3 dose extended schedule (0-6-18 months) for the HPV vaccine Gardasil-9 provide similar immune responses and short term protection against HPV infection compared to the regular 3 dose schedule (0-2-6 months) in high risk women in Vietnam

DETAILED DESCRIPTION:
Primary objective:

To determine whether antibody geometric mean titer (GMT) to vaccine type HPV16 and HPV18 at 7 months (m) are non-inferior between female sex workers (FSW) aged 18-26 years who received the standard (0, 2m, 6m) and those received the extended 3-dose (at 0, 6m and 18m) 9vHPV schedule and age-matched non-FSW who received an extended 3-dose (at 0, 6m and 18m) 9vHPV schedule. This extended 3-dose schedule is in line with the recommended schedule by the vaccine manufacturer in Vietnam.

Secondary objectives:

1. To compare antibody GMT at 2m, 7m, 18m and 19m between FSW who are HPV DNA+/seropositive with FSW who are HPV DNA-/seronegative at baseline.
2. To compare antibody GMT at 18m and 19m between FSW and non-FSW.
3. To determine cellular immune responses to HPV16 and 18 at baseline, 2m, 7m, 18m and 19m.
4. To measure incidence and 6m/12m/18m persistent HPV infection.

Primary hypothesis:

HPV antibody GMT to HPV16 and 18 in FSW is non-inferior to those of young women of the same age group (non-FSW) at 7m.

Secondary hypothesis:

1. HPV antibody GMT are similar at 2m, 7m, 18m and 19m between FSW who are HPV DNA+/seropositive and HPV DNA-/seronegative at month 0.
2. HPV antibody GMT are similar at 18m and 19m between FSW and non-FSW who received the extended schedule.
3. Cellular immune responses to HPV16 and 18 are similar between FSW and non-FSW at 2m, 7m, 18m and 19m who received the extended schedule.
4. No new vaccine-type HPV infection in FSW and non-FSW in all groups at 6m, 12m, 18m.

ELIGIBILITY:
Inclusion Criteria:

* Is between the reporting ages of 18-26 years at the time of recruitment.
* Engage in commercial sex in the last 6m (for FSW group) or have engaged in sexual activity (non-FSWs)
* Willing and able to give written informed consent.
* Willing to complete the follow-up requirements of the study.

Exclusion criteria

Participants meeting any of the following criteria will be excluded from the trial:

* Pregnant or possibly pregnant
* Has received any HPV vaccine previously
* Has an axillary temperate greater than 38°C
* Known allergies to any vaccine component
* incapacity to provide consent
* Currently receiving immunosuppressive medication or anti-cancer chemotherapy.
* Known HIV infection.
* Known Congenital immune deficiency syndrome.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female sex workers or female non-sex workers aged 18-26 years
Enrollment: 300 (Estimated)
Dates: Start 2024-12-14 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison between antibody responses after the 3rd dose ofregular vaccine schedules among FSW and after the 2nd dose of the extended schedule | 7 months from the first doses
  geometric mean titer (GMT) ratios and 95% confidence intervals (CI) of HPV- specific antibody responses to HPV16 and HPV18 at 7m between FSWs aged 18-26 years who received either the standard (0, 2m, 6m) or extended 3-dose (at 0, 6m and 18m) 3-dose 9vHPV schedule and age-matched non-FSWs who received the extended 3-dose 9vHPV schedule (at 0, 6m and 18m).

SECONDARY OUTCOMES:
Comparison of antibody responses after each doses among FSW according to HPV infection status pre-vaccination | 19 months after the 1st doses
  Antibody GMT at 2m, 7m, 18m and 19m between FSW who are HPV DNA+/seropositive with FSW who are HPV DNA-/seronegative at baseline.
Comparison of antibody response after 3 doses of extended schedule between FSW and non-FSW | 19 month after the first doses
  Antibody GMT at 18m and 19m between FSW and non-FSW.
Celular response after each vaccine dose | 19 months after the 1st dose
  Proportion of HPV16 and 18-specific B/T cells at baseline, 2m, 7m, 18m and 19m.
HPV persistent during 19 month or more among vaccines | at least 19 months after the first dose
  4. Incidence (detection of the specific-type HPV DNA at least once during the follow-up period) and persistent HPV infection (defined as detection of the same HPV type in at least 2 samples not interrupted by negative sample during the follow-up period).

CONTACTS AND LOCATIONS:
Overall Officials: Hong T Duong, MD, PhD, Study Director — National Institute of Hygiene and Epidemiology, Vietnam; Trang V Nguyen, PhD, Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam; Tuan A Le, MD, PhD, Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam
Locations (3):
- Murdoch Children Research Institute, Parkville, Victoria, Australia
- Vietnam (2):
  - Center for Supporting Community Development Initiatives SCDI-Vietnam, Haiphong
  - Hai Phong Center for Disease Control, Haiphong

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Results will be reported as grouped data

REFERENCES:
- [Background] Nguyen TP, Luu HN, Nguyen MVT, Tran MT, Tuong TTV, Tran CTD, Boffetta P. Attributable Causes of Cancer in Vietnam. JCO Glob Oncol. 2020 Feb;6:195-204. doi: 10.1200/JGO.19.00239. PMID 32045545
- [Background] Thi Nguyen DN, Simms K, Vu Nguyen HQ, Van Tran T, Nguyen NH, LaMontagne DS, Castle P, Canfell K. The burden of cervical cancer in Vietnam: Synthesis of the evidence. Cancer Epidemiol. 2019 Apr;59:83-103. doi: 10.1016/j.canep.2018.11.008. Epub 2019 Jan 30. PMID 30710841
- [Background] Vandepitte J, Lyerla R, Dallabetta G, Crabbe F, Alary M, Buve A. Estimates of the number of female sex workers in different regions of the world. Sex Transm Infect. 2006 Jun;82 Suppl 3(Suppl 3):iii18-25. doi: 10.1136/sti.2006.020081. PMID 16735288
- [Result] VAN Trang N, Prem K, Toh ZQ, Viet Ha BT, Ngoc Lan PT, Tran HP, Pham QD, VAN Khuu N, Jit M, Luu DT, Khanh Ly LT, Cao V, LE-Ha TD, Bright K, Garland SM, Anh DD, Mulholland K. Prevalence and Determinants of Vaginal Infection With Human Papillomavirus Among Female University Students in Vietnam. In Vivo. 2022 Jan-Feb;36(1):241-250. doi: 10.21873/invivo.12697. PMID 34972721
- [Result] Tuan LA, Prem K, Pham QD, Toh ZQ, Tran HP, Nguyen PD, Mai CTN, Ly LTK, Cao V, Le-Ha TD, Tuan NA, Jit M, Bright K, Brisson M, Nguyen TV, Garland S, Anh DD, Trang NV, Mulholland K. Anal human papillomavirus prevalence and risk factors among men who have sex with men in Vietnam. Int J Infect Dis. 2021 Nov;112:136-143. doi: 10.1016/j.ijid.2021.09.016. Epub 2021 Sep 10. PMID 34517047
- [Result] Pham QD, Prem K, Le TA, Van Trang N, Jit M, Nguyen TA, Cao V, Le-Ha TD, Chu MTN, Le LTK, Toh ZQ, Brisson M, Garland S, Murray G, Bright K, Dang DA, Tran HP, Mulholland EK. Prevalence and risk factors for human papillomavirus infection among female sex workers in Hanoi and Ho Chi Minh City, Viet Nam: a cross-sectional study. Western Pac Surveill Response J. 2022 Nov 7;13(4):1-11. doi: 10.5365/wpsar.2022.13.4.894. eCollection 2022 Oct-Dec. PMID 36817494
- [Result] Hernandez BY, Vu Nguyen T. Cervical human papillomavirus infection among female sex workers in southern Vietnam. Infect Agent Cancer. 2008 Apr 23;3:7. doi: 10.1186/1750-9378-3-7. PMID 18433504
- [Result] Brown B, Blas M, Cabral A, Carcamo C, Gravitt P, Halsey N. Randomized trial of HPV4 vaccine assessing the response to HPV4 vaccine in two schedules among Peruvian female sex workers. Vaccine. 2012 Mar 16;30(13):2309-14. doi: 10.1016/j.vaccine.2012.01.058. Epub 2012 Feb 1. PMID 22306855
- [Result] Dobson SR, McNeil S, Dionne M, Dawar M, Ogilvie G, Krajden M, Sauvageau C, Scheifele DW, Kollmann TR, Halperin SA, Langley JM, Bettinger JA, Singer J, Money D, Miller D, Naus M, Marra F, Young E. Immunogenicity of 2 doses of HPV vaccine in younger adolescents vs 3 doses in young women: a randomized clinical trial. JAMA. 2013 May 1;309(17):1793-802. doi: 10.1001/jama.2013.1625. PMID 23632723